CLINICAL TRIAL: NCT03403218
Title: Translation and Validation of the Spanish Version of the BESTest and Mini-BESTest
Brief Title: Spanish Version of the Balance Evaluation Systems Test and Mini Balance Evaluation Systems Test
Acronym: BESTest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Instituto Aragones de Ciencias de la Salud (Other Government)
Responsible Party: Principal Investigator, Pilar Dominguez-Olivan, PhD. Titular de Universidad., Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI17/0282
Record Dates: First submitted 2017-09-23; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Balance
Keywords: balance, risk of falling
MeSH Terms: interventions — Diagnosis-Related Groups

STUDY DESIGN:
Intervention Model Description: single group assignment. cross-sectional survey.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- case group (Experimental): BESTest, mini-BESTest, Berg scale and FES (falls efficacy scale) (in Spanish version is administrated in case group.
  Interventions: Behavioral: Case group

INTERVENTIONS:
Behavioral: Case group — assessment of quality on posture, transfers and displacement

SUMMARY:
This study aim to translate the BESTest and mini-BESTest to Spanish, adapt it and investigate its validity in spanish population.

DETAILED DESCRIPTION:
To translate the BESTest and mini-BESTest to Spanish, adapt it and investigate its validity in spanish. Check its metric properties in relation to other balance tests.

ELIGIBILITY:
Inclusion Criteria: healthy subjects without diagnosed balance problems.

-

Exclusion Criteria:

* Diagnosed balance problems.
* One falling in the last three months.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Concurrent validity of Best test- 1 | 1 month
  concurrent validity of BESTest compare to other model balance tests

SECONDARY OUTCOMES:
Psychometric properties of Spanish version of BESTest. | 1 year
  To perform a detailed analysis of the psychometric properties of the BESTest Spanish version.
Psychometric properties of Spanish version of mini-BESTest. | 1 year
  To perform a detailed analysis of the psychometric properties of the mini-BESTest Spanish version.

OTHER OUTCOMES:
concurrent validity of mini-BESTest | 1 month
  concurrent validity of mini-BESTest compare to Berg scale and FES.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Mr Lanas-Arbeloa, Study Chair — Instituto de Investigacion Sanitaria de Aragon
Locations (1):
- Facultad de Ciencias de la Salud, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Blind date analysis researcher. By coding affiliation information.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: data will become available from October 2017 and for three months.
Access Criteria: affiliation date are code. The rest of registration is shared.

REFERENCES:
- [Derived] Dominguez-Olivan P, Gasch-Gallen A, Aguas-Garcia E, Bengoetxea A. Validity and reliability testing of the Spanish version of the BESTest and mini-BESTest in healthy community-dwelling elderly. BMC Geriatr. 2020 Nov 4;20(1):444. doi: 10.1186/s12877-020-01724-3. PMID 33148216

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-09-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT03403218/SAP_000.pdf
  • Informed Consent Form (2017-09-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT03403218/ICF_001.pdf
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT03403218/Prot_002.pdf